CLINICAL TRIAL: NCT05990777
Title: Assessment of Knowledge and Attitude Toward Obstructive Sleep Apnea in Medical Teams: Multicenter Study
Brief Title: Assessment of Knowledge and Attitude Toward Obstructive Sleep Apnea in Medical Teams
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU22-1
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: OSA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea (OSA) is a serious and often underreported condition, despite its highly prevalent distribution. Medical teams play an integral role in screening and managing patients with a high risk of developing OSA.

ELIGIBILITY:
Inclusion Criteria:

Medical teams including:

* Students of medical schools and dentistry
* General practitioners
* Dentists
* Medical specialists
* Highly trained nurses (HIN)

Exclusion Criteria:

* Non- medical personnel's

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical teams including:
  All responders to the questionnaires will be included regarding that they belong to these groups- within the study period
  * Students of medical schools and dentistry
  * General practitioners
  * Dentists
  * Medical specialists
  * Highly trained nurses (HIN)
Sampling Method: Non-Probability Sample
Enrollment: 377 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
explores the knowledge and attitude towards OSA among medical teams | 3 months
  frequency

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Aliae AR Mohamed-Hussein, Asyut
  - Aliae Mohamed-Hussein, Asyut

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request